CLINICAL TRIAL: NCT06539754
Title: Patient Satisfaction of the Environment During Cesarean Delivery
Brief Title: Patient Satisfaction During Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-0158
Record Dates: First submitted 2024-07-08; First posted 2024-08-06 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Patient Satisfaction
Keywords: Cesarean delivery
MeSH Terms: conditions — Patient Satisfaction | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized in 1:1 stratification to receive music during their procedure or not. Participants will not be aware of the intervention. If a patient is randomized into music, they will be offered headphones to listen to during their procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No music (No Intervention): Participants who undergo cesarean delivery will not have music available to listen to during the procedure.
- Music (Experimental): Participants who undergo cesarean delivery will have music of their choice played through bone conduction headphones.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Participants will have bone conducting headphones available to listen to the music of their choice from premade Spotify playlists.
  Arms: Music

SUMMARY:
The goal of this interventional study is to determine whether the option to listen to music during cesarean delivery increases the participants satisfaction. Participants and their support person will be asked to fill out a short survey and mark their satisfaction on a visual analog scale. Vital signs will be recorded during their procedure.

DETAILED DESCRIPTION:
Currently, our institution does not routinely offer music during cesarean delivery. The goal of this study would be to determine whether the option to listen to music improves patient satisfaction. Also, the study would examine support person satisfaction and changes in maternal vital signs from prior to entering the operating room as compared to prior to exiting the operating room in a sample of patients. If positive satisfaction results are noted in those randomized to the music arm, this would be a low-cost intervention that providers could utilize to increase patient satisfaction during surgery.

This will be a prospective randomized controlled trial to determine whether the option of music being played in the operating room can impact the experience for the patient. Subjects will be randomized via central computer-generated randomization 1:1 to either have music played during their procedure or no music played during their procedure. A per protocol analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Second or third cesarean delivery
* Scheduled cesarean delivery at Geisinger Medical Center
* Able and willing to provide consent
* English speaking
* Greater than or equal to 37 weeks' gestation

Exclusion Criteria:

* Fetal anomaly
* Multifetal gestation
* Hearing loss requiring a sign interpreter or hearing aids
* Planned general anesthesia
* Intrauterine fetal demise
* Participants that present in labor or require urgent/emergent cesarean delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction | This is collected during the study duration, on average 6 hours.
  Visual analog scales from 0-10 (0=extremely unsatisfied, 10=extremely satisfied) will be collected by the patient marking on the line prior to the procedure and during skin closure.

SECONDARY OUTCOMES:
Support person satisfaction | This is collected through the duration of the study, on average 6 hours,
  Visual analog scales from 0-10 (0=extremely unsatisfied, 10=extremely satisfied) will be collected by the support person marking on a line during the participant's skin closure.
Heart rate | This will be collected during the study duration, an average 6 hours.
  Participants heart rate will be recorded at the time of consent and during skin closure.
Music and satisfaction | This is collected during the study duration, on average 6 hours.
  Patient's will be asked after their procedure whether they believe music did or would have improved their satisfaction during cesarean delivery using a visual analog scale (0-10)
Blood pressure | This will be collected during the study duration, an average 6 hours.
  Participants blood pressure (systolic and diastolic) will be recorded at the time of consent and during skin closure.

CONTACTS AND LOCATIONS:
Overall Officials: Awathif D Mackeen, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No personal or identifying information from individual participants will be collected. Aggregate data will thus be reported.